CLINICAL TRIAL: NCT01484327
Title: Multicentre, Open-label, Non-interventional Observational Clinical Study Lasting 48 Weeks in Patients With Heart Failure or Reduced Left Ventricular Ejection Fraction Following Acute Myocardial Infarction Who Are Treated With Carvedilol
Brief Title: Carvedilol Vascular Efficacy Trial
Acronym: CARVEDIA
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008-CAR-EL-02; Carvedia - 02 (Other: Elpen Pharmaceutical Co Inc)
Record Dates: First submitted 2011-11-23; First posted 2011-12-02 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2011-11

CONDITIONS: Heart Failure; Acute Myocardial Infarction
Keywords: Heart Failure; Acute Myocardial Infarction; LVEF
MeSH Terms: conditions — Heart Failure | interventions — Carvedilol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carvedilol, LVEF, Heart Failure: Patients with Heart Failure on carvedilol therapy measured for their LVEF value
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Minimum dosage 3.125 mg Χ 2, Maximum dosage 50 mg
  Other Names: Carvepen

SUMMARY:
Beta-blockers should be administered to all patients with heart failure stages II to IV NYHA. It should also be administered to patients with stage I after myocardial infarction. The low ejection fraction, especially after myocardial infarction is a strong indication for beta-blockers, as many studies indicate that administration of these drugs substantially reduces cardiovascular mortality. Beta-blockers reduce mortality and hospitalizations and improve the operational phase for all categories of patients with heart failure. Since beta-blockers, only carvedilol, metoprolol, and recently visoprololi nevimpololi have shown these benefits and thus, only those have to be administered.

The clinical study Carvedia aims to observe and record the action of beta-blocker carvedilol on cardiac function in patients with heart failure or reduced left ventricular ejection fraction after acute myocardial infarction.

DETAILED DESCRIPTION:
The relationship between stroke volume, which is extruded from the left ventricle gives a measure for the restrictive left ventricular function. Any patient with known cardiovascular disease should undergo assessment of left ventricular function by measuring the ejection fraction. Several studies have shown that when the ejection fraction (LVEF), which measures the heart's ability to eject blood to the aorta does not exceed 40% (natural price ^ 50%) increased dramatically in the post-infarction mortality. The ejection fraction as a reliable predictor, can be measured by ultrasonography. The reduced ejection fraction is associated with an increased risk of life-threatening arrhythmias, heart failure and death. The low ejection fraction, especially after myocardial infarction is a strong indication for beta-blockers, as many studies indicate that administration of these drugs substantially reduces cardiovascular mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients visiting outpatient clinics.
2. Male or female patients over 18 years
3. Patients with mild heart failure and history of symptoms according to the instructions of the European Society of Cardiology (ESC)
4. Patients who entered the study have LVEF <40% in echocardiography
5. Patients with new diagnosis of heart failure
6. Patients who have left ventricular ejection fraction after acute myocardial infarction <40%
7. Patients who have been treated in hospital during the previous month before their inclusion in the study
8. Patients who have signed the consent form for recording and processing of personal data.
9. Patients who are willing to comply with the requirements of the study
10. Patients who are treated with carvedilol for at least a month before their inclusion in this

Exclusion Criteria:

1. Patients under 18 years
2. Patients with unstable chronic heart failure
3. Patients with unstable hemodynamic profiles
4. Patients with heart valve disease
5. Patients with hypertrophic cardiomyopathy
6. Patients with unstable angina or active myocarditis
7. Patients with contraindications to treatment with beta-adrenergic receptors
8. Patients who have not consented to recording and processing of personal the data.
9. Women pregnant or breastfeeding
10. Patients have been treated in hospital during the preceding months before their inclusion in the study
11. Patients treated with carvedilol for less than one month

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Heart Failure and post-MI LVEF<40%
Sampling Method: Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction LVEF(%) | 0 (baseline), 48 weeks (12 months)
  Change from baseline in Left Ventricular Ejection Fraction LVEF(%) at 12 months.

SECONDARY OUTCOMES:
Number of study participants with Adverse Events | 0 (baseline), 24 weeks (6 months), 48 weeks (12 months)
  Safety of carvedilol administration (reported AEs) from baseline until 12 months of treatment.
Cardedilol dosage range | 0 (baseline), 24 weeks (6 months), 48 weeks
  Relation between carvedilol dose titration and change in LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Tziakas, A Professor, Principal Investigator — University General Hospital of Alexandroupolis, Cardiology Department
Locations (1):
- Cardiology University Clinic, Alexandroupoli, Greece

REFERENCES:
- See also: 13th national congress for heart failure (Hellenic Society of Heart Failure) — http://heartfailuregreece.blogspot.com/2012/02/13.html
- See also: European Society of Cardilogy - Heart Failure Congress 2012, Belgrade, Abstract No 60343 — http://escol.escardio.org/MyESC/modules/congress/Abstract/default.aspx?eventID=156